CLINICAL TRIAL: NCT04817527
Title: Edaravone Dexborneol for Treatment of Acute Ischemic Stroke With Endovascular Therapy in Extended Time Windows (EXISTENT):a Prospective, Randomized, Open-label, Multi-centre Study
Brief Title: Edaravone Dexborneol for Treatment of Acute Ischemic Stroke With Endovascular Therapy in Extended Time Windows
Acronym: EXISTENT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJTU1AF2021LSK-065
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2021-08

CONDITIONS: Stroke, Ischemic
Keywords: Endovascular therapy; Extended Time Windows
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Edaravone Dexborneol (Experimental)
  Interventions: Drug: Edaravone Dexborneol
- conventional therapy (No Intervention): conventional therapy of acute ischemic stroke after Endovascular Therapy based on Chinese guidelines for endovascular therapy

INTERVENTIONS:
Drug: Edaravone Dexborneol — Intravenous injections of edaravone dexborneol (37.5mg in 0·9% NaCl) BID for 7-14days.
  Arms: Edaravone Dexborneol

SUMMARY:
To explore the safety and efficacy of edaravone dexborneol for patients of acute ischemic stroke received endovascular therapy in extended time windows.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 years of age;
2. Acute ischemic stroke with National Institute of Health Stroke Scale (NIHSS) ≥ 10 and Volume of infarction on DWI <31ml or with a NIHSS ≥20 and 31ml<Volume of infarction<51ml(DWI);
3. Patients who presented with acute ischemic stroke and a large vessel occlusion in the anterior circulation;
4. Endovascular Therapy in 6-24 hours of stroke onset;
5. The availability of informed consent.

Exclusion Criteria:

1. First ever stroke or mRS≤1 after previous disease;
2. Hemorrhagic stroke: cerebral hemorrhage, subarachnoid hemorrhage;
3. Coagulation disorders, systematic hemorrhagic tendency, thrombocytopenia
4. Severe hepatic or renal dysfunction, increase in ALT or AST (more than 2 times of upper limit of normal value), increase in serum creatinine (more than 1.5 times of upper limit of normal value) or requiring dialysis;
5. Severe cardiac or pulmonary disease;
6. Patients with malignant tumor or under antineoplastic therapy with estimated lifetime less than 3 months;
7. Pregnancy, plan to get pregnant or during lactation;
8. Patients with contraindication or allergic to any ingredient of drugs in our study;
9. Unsuitable for this clinical studies assessed by researcher

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with modified Rankin Score 0 to 3 on day 90 | 90 days
Proportion of symptomatic intracranial hemorrhage (sICH) | 48 hours
mTICI grade (<2 b、≥2 b) stratified for primary outcome analysis | 90 days

SECONDARY OUTCOMES:
Changes in National Institute of Health stroke scale (NIHSS) on day 2,7,14 | 14 days
Distribution of modified Rankin Score after the treatment | 90 days
Change in infarct volume | 7 days
The proportion of patients with Barthel Index (BI) score greater than or equal to 95 on day 14, 30, 90 | 90 days
Activity of Daily Living Scale(ADL) score on day 14, 30, 90 | 90 days
Montreal Cognitive Assessment(MoCA) score on day 14, 30, 90 | 90 days
Serum inflammatory factors changes on day 1 and day 7 | 7 days
Proportion of PH1 and PH2 within 48 hours after the treatment | 48 hours
Midline shift on the CT scan | 7 days
Proportion of death due to any cause | 90 days
Proportion of Serious adverse events(SAE) | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No